CLINICAL TRIAL: NCT01865773
Title: Role of HFR Cartridge in the Removal of Mediators of Inflammation and P-cresol in Hemodialysis Patients
Brief Title: HFR Cartridge and Inflammation
Acronym: HFR
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Federico II University (Other)
Responsible Party: Principal Investigator, Eleonora Riccio, MD, Federico II University
Allocation: Not Applicable | Model: Single Group | Masking: None
Other Study IDs: HFR13; HFRinflamm
Record Dates: First submitted 2013-05-23; First posted 2013-05-31 (Estimated); Last update posted 2013-05-31 (Estimated); Status verified 2013-04

CONDITIONS: Inflammatory Status; P-cresol

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- HFR (Experimental): We selected 8 inflamed chronic HD patients, which underwent a single 240 minutes HFR session
  Interventions: Procedure: HFR dialysis

INTERVENTIONS:
Procedure: HFR dialysis — HFR is a dialysis technique that combines the processes of diffusion, convection and adsorption. In this double chamber hemodiafiltration system, the ultrafiltrate is reinfused after its passage (and opportune modification) through a resin cartridge.
  Other Names: hmodiafiltration with on line reinfusion of ultrafiltrate

SUMMARY:
A major limitation of standard hemodialysis is that it does not clear the plasma from interleukin-6 (IL-6) and p-cresol, two uremic toxins responsible for the high cardiovascular risk in end stage renal disease (ESRD). In the present study, we evaluated whether these compounds are removed by HFR-Supra, a double-chamber hemodiafiltration system in which the ultrafiltrate (UF) returns to the patient after its regeneration through a resin cartridge. We selected 8 inflamed chronic hemodialysis (HD) patients, which underwent a single 240 minutes HFR session. We studied the change in both IL-6 and p-cresol circulating levels, by comparing pre- and post-HFR serum concentrations. In addition, we compared Il-6 and p-cresol levels in the UF entering (UFin) and exiting (UFout) from the cartridge, either at the start or at the end of the HFR session. The proinflammatory activity of UFin and UFout was determined by evaluating the changes that they induced in IL-6 messenger ribonucleic acid (mRNA) expression and release in peripheral blood mononuclear cells (PBMC) collected from 8 healthy volunteers and cultured in vitro for 24 hr.

ELIGIBILITY:
Inclusion Criteria:

* HD patients undergoing three weekly haemodialysis > 1 year

Exclusion Criteria:

* none

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 8 (Actual)
Dates: Start 2011-01; Primary Completion 2012-04 (Actual); Study Completion 2012-09 (Actual)

PRIMARY OUTCOMES:
IL-6 removal by a single session of HFR-Supra | The evaluation will be performed for the duration of a single HFR session of 240 minutes
  We studied the change in IL-6 circulating levels, by comparing pre- and post-HFR serum concentrations. In addition, we compared IL-6 levels in the UF entering (UFin) and exiting (UFout) from the cartridge, either at the start or at the end of the HFR session. The proinflammatory activity of UFin and UFout was determined by evaluating the changes that they induced in IL-6 mRNA expression and release in peripheral blood mononuclear cells (PBMC) collected from 8 healthy volunteers and cultured in vitro for 24 hr.
P-cresol removal by a single HFR session | The evaluation will be performed for the duration of a single HFR session of 240 minutes
  We studied the change in p-cresol circulating levels, by comparing pre- and post-HFR serum concentrations. In addition, we compared p-cresol levels in the UF entering (UFin) and exiting (UFout) from the cartridge, either at the start or at the end of the HFR session.

CONTACTS AND LOCATIONS:
Locations (1):
- federico II university, department of nephrology, Naples, Naples, Italy

REFERENCES:
- [Derived] Riccio E, Cataldi M, Minco M, Argentino G, Russo R, Brancaccio S, Memoli A, Grumetto L, Postiglione L, Guida B, Memoli B. Evidence that p-cresol and IL-6 are adsorbed by the HFR cartridge: towards a new strategy to decrease systemic inflammation in dialyzed patients? PLoS One. 2014 Apr 22;9(4):e95811. doi: 10.1371/journal.pone.0095811. eCollection 2014. PMID 24755610